CLINICAL TRIAL: NCT06816381
Title: Characterizing Uterine and Ovarian Tissue Stiffness Via Shear Wave Elastography in Non-Infertile, Fertile, and Infertile Women with Normal Anatomy Across the Menstrual Cycle: a Pilot Study
Brief Title: Quantifying Uterine Elastography in Menstruating Women
Acronym: QUEST
Status: Recruiting | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: 2401-BRG-003-FB
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Infertility (IVF Patients); Infertility Assisted Reproductive Technology
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples obtained from participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Nulliparous Women with No Known infertility: Female patients with normal menstrual cycles, normal ovarian and uterine anatomy and with no known prior pregnancy (including miscarriages, terminations, ectopic pregnancies, preterm and full term deliveries)
  Interventions: Device: Shear wave elastography measurements
- Gravid Women with No Known infertility: Female patients with normal menstrual cycles, normal ovarian and uterine anatomy with at least one prior full term vaginal delivery with no known infertility
  Interventions: Device: Shear wave elastography measurements
- Primary Infertile Women Without Uterine Factor Infertility: Female patients with normal menstrual cycles, normal ovarian and uterine anatomy and with no known prior pregnancy (including miscarriages, terminations, ectopic pregnancies, preterm and full term deliveries) that has been diagnosed with primary infertility
  Interventions: Device: Shear wave elastography measurements

INTERVENTIONS:
Device: Shear wave elastography measurements — Shear wave elastography measurements in kilopascals via ultrasound

SUMMARY:
This study is aiming to characterize the elasticity of the female reproductive tract including the uterus, cervix and ovary using shear wave elastography at different times during the menstrual cycle and define the standard reference range of normal uterine and ovarian elasticity. By doing so, the potential of using shear wave elastography to diagnose and predict outcomes for patients seeking fertility treatment might be established.

ELIGIBILITY:
Group A

Inclusion Criteria:

* Patients with normal menstrual cycles lasting 28-34 days
* Patients with normal uterine anatomy
* Patients with no prior pregnancy history including miscarriages, terminations, ectopic pregnancies, preterm deliveries, or full-term deliveries
* Patient who have no known infertility (i.e. women who have not tried to conceive)

Exclusion Criteria:

* BMI ≥ 35
* Current use of intrauterine devices (IUDs), hormonal implants, or hormonal birth control medications. Participants on hormonal birth control interested in study participation may be included following one month of discontinuation of hormonal medication.
* History of uterine surgery (i.e hysteroscopy, dilation and curettage, myomectomy)
* History of ovarian surgery (i.e ovarian cystectomy, oophorectomy, removal of -endometrioma)
* History of surgically-confirmed or clinically suspected endometriosis or ultrasound evidence of endometriosis (i.e endometrioma)
* Currently present or surgically corrected uterine anomalies
* Ultrasound evidence of or history of communicating hydrosalpinx
* Ultrasound evidence of or history of leiomyomas
* Ultrasound evidence of adenomyosis based on the Morphological Uterus Sonographic Assessment criteria (MUSA) (19)
* Ultrasound evidence of ovarian pathology including mature teratoma/dermoid cyst, persistent functional cysts larger than 2 cm, or ovarian cancer.

Group B

Inclusion Criteria:

* Patients with normal menstrual cycles lasting 28 days to 34 days.
* Patients with normal uterine and ovarian anatomy (absence of gross pathology on screening visit ultrasound)
* Patients with at least one prior full-term vaginal delivery with time to conception less than one year without the use of assisted reproductive technology.

Exclusion Criteria

* BMI ≥ 35
* Current use of intrauterine devices (IUDs), hormonal implants, or hormonal birth control medications. Participants on hormonal birth control interested in study participation may be included following one month of discontinuation of hormonal medication.
* History of cesarean section
* Patient who have no known secondary infertility (i.e. women who have not tried to conceive)
* Diagnosis of secondary infertility (i.e women who have attempted pregnancy for 12 months without success)
* History of uterine surgery (i.e hysteroscopy, dilation and curettage, myomectomy)
* History of ovarian surgery (i.e ovarian cystectomy, oophorectomy, removal of endometrioma)
* History of surgically-confirmed or clinically suspected endometriosis or ultrasound evidence of endometriosis (i.e endometrioma)
* Currently present or surgically corrected uterine anomalies
* Ultrasound evidence of or history of communicating hydrosalpinx
* Ultrasound evidence of or history of leiomyomas
* Ultrasound evidence of adenomyosis based on the Morphological Uterus Sonographic Assessment criteria (MUSA) (19)
* Ultrasound evidence of ovarian pathology including mature teratoma/dermoid cyst, persistent functional cysts larger than 2 cm, or ovarian cancer.

Group C

Inclusion Criteria:

* Patients with normal menstrual cycles lasting 28 days to 34 days.
* Patients with normal uterine and ovarian anatomy (absence of gross pathology on screening visit ultrasound)
* Patient with no prior pregnancy history including miscarriages, terminations, ectopic pregnancies, preterm deliveries, or full-term deliveries (i.e gravity equals zero).
* Patient with diagnosis of primary infertility, with attempted conception for at least 12 months if younger than 35 years and attempted conception for at least 6 months if 35 years or older.

Exclusion Criteria

* BMI ≥ 35
* Current use of intrauterine devices (IUDs), hormonal implants, or hormonal birth control medications. Participants on hormonal birth control interested in study participation may be included following one month of discontinuation of hormonal medication.
* History of three or more failed euploid embryo transfers
* Severe male factor infertility including severe oligozoospermia and cryptozoospermia
* History of uterine surgery (i.e hysteroscopy, dilation and curettage, myomectomy)
* History of ovarian surgery (i.e ovarian cystectomy, oophorectomy, removal of endometrioma)
* History of surgically-confirmed or clinically suspected endometriosis or ultrasound evidence of endometriosis (i.e endometrioma)
* Currently present or surgically corrected uterine anomalies
* Ultrasound evidence of or history of communicating hydrosalpinx
* Ultrasound evidence of or history of leiomyomas
* Ultrasound evidence of adenomyosis based on the Morphological Uterus Sonographic Assessment criteria (MUSA) (19)
* Ultrasound evidence of ovarian pathology including mature teratoma/dermoid cyst, persistent functional cysts larger than 2 cm, or ovarian cancer.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Nulliparous women with no known infertility, gravid women with no known infertility and primary infertile women without uterine factor infertility
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Shear wave elastography parameters | 3-4 months from enrollment
  shear wave elastography measurements in kilopascals

CONTACTS AND LOCATIONS:
Locations (1):
- RMA, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 6. https://www.sart.org/patients/a-patients-guide-to-assisted-reproductive-technology/general-information/success-rates/
- [Background] Vora Z, Manchanda S, Sharma R, Das CJ, Hari S, Mathur S, Kumar S, Kachhawa G, Khan MA. Transvaginal Shear Wave Elastography for Assessment of Endometrial and Subendometrial Pathologies: A Prospective Pilot Study. J Ultrasound Med. 2022 Jan;41(1):61-70. doi: 10.1002/jum.15679. Epub 2021 Mar 1. PMID 33645765
- [Background] Shao J, Shi G, Qi Z, Zheng J, Chen S. Advancements in the Application of Ultrasound Elastography in the Cervix. Ultrasound Med Biol. 2021 Aug;47(8):2048-2063. doi: 10.1016/j.ultrasmedbio.2021.04.009. Epub 2021 May 26. PMID 34049726
- [Background] Van den Bosch T, de Bruijn AM, de Leeuw RA, Dueholm M, Exacoustos C, Valentin L, Bourne T, Timmerman D, Huirne JAF. Sonographic classification and reporting system for diagnosing adenomyosis. Ultrasound Obstet Gynecol. 2019 May;53(5):576-582. doi: 10.1002/uog.19096. No abstract available. PMID 29790217
- [Background] Soliman AA, Wojcinski S, Degenhardt F. Ultrasonographic examination of the endometrium and myometrium using acoustic radiation force impulse (ARFI) imaging technology: An initial experience with a new method. Clin Hemorheol Microcirc. 2015;59(3):235-43. doi: 10.3233/CH-141842. PMID 24840338
- [Background] Kabukcu C, Cabus U, Oztekin O, Fenkci V. The strain rate of endometrium measured by real-time sonoelastography as a predictive marker for pregnancy in gonadotropin stimulated intrauterine insemination cycles. J Obstet Gynaecol Res. 2021 Oct;47(10):3561-3570. doi: 10.1111/jog.14921. Epub 2021 Jul 12. PMID 34254413
- [Background] Batur A, Yavuz A, Ozgokce M, Bora A, Bulut MD, Arslan H, Alpaslan M. The utility of ultrasound elastography in differentiation of endometriomas and hemorrhagic ovarian cysts. J Med Ultrason (2001). 2016 Jul;43(3):395-400. doi: 10.1007/s10396-016-0701-5. Epub 2016 Feb 15. PMID 26880060
- [Background] Swierkowski-Blanchard N, Boitrelle F, Alter L, Selva J, Quibel T, Torre A. Uterine contractility and elastography as prognostic factors for pregnancy after intrauterine insemination. Fertil Steril. 2017 Apr;107(4):961-968.e3. doi: 10.1016/j.fertnstert.2017.02.002. Epub 2017 Mar 7. PMID 28283264
- [Background] Altunkeser A, Inal ZO, Baran N. Evaluation of Ovaries in Patients with Polycystic Ovary Syndrome using Shear Wave Elastography. Curr Med Imaging. 2020;16(5):578-583. doi: 10.2174/1573405615666190114150538. PMID 32484092
- [Background] Raga F, Bonilla-Musoles F, Casan EM, Klein O, Bonilla F. Assessment of endometrial volume by three-dimensional ultrasound prior to embryo transfer: clues to endometrial receptivity. Hum Reprod. 1999 Nov;14(11):2851-4. doi: 10.1093/humrep/14.11.2851. PMID 10548635
- [Background] Barrett F, Willson S, Werner M. Advancements in the application of uterine ultrasound elastography. Curr Opin Obstet Gynecol. 2024 Jun 1;36(3):181-185. doi: 10.1097/GCO.0000000000000949. Epub 2024 Mar 26. PMID 38656810
- [Background] Hawkins Bressler L, Steiner A. Anti-Mullerian hormone as a predictor of reproductive potential. Curr Opin Endocrinol Diabetes Obes. 2018 Dec;25(6):385-390. doi: 10.1097/MED.0000000000000440. PMID 30299431
- [Background] Zaniker EJ, Zhang M, Hughes L, La Follette L, Atazhanova T, Trofimchuk A, Babayev E, Duncan FE. Shear wave elastography to assess stiffness of the human ovary and other reproductive tissues across the reproductive lifespan in health and diseasedagger. Biol Reprod. 2024 Jun 12;110(6):1100-1114. doi: 10.1093/biolre/ioae050. PMID 38609185
- [Background] Cedars MI. Evaluation of Female Fertility-AMH and Ovarian Reserve Testing. J Clin Endocrinol Metab. 2022 May 17;107(6):1510-1519. doi: 10.1210/clinem/dgac039. PMID 35100616
- [Background] Scott RT Jr, Upham KM, Forman EJ, Hong KH, Scott KL, Taylor D, Tao X, Treff NR. Blastocyst biopsy with comprehensive chromosome screening and fresh embryo transfer significantly increases in vitro fertilization implantation and delivery rates: a randomized controlled trial. Fertil Steril. 2013 Sep;100(3):697-703. doi: 10.1016/j.fertnstert.2013.04.035. Epub 2013 Jun 1. PMID 23731996
- [Background] Scott RT Jr, Ferry K, Su J, Tao X, Scott K, Treff NR. Comprehensive chromosome screening is highly predictive of the reproductive potential of human embryos: a prospective, blinded, nonselection study. Fertil Steril. 2012 Apr;97(4):870-5. doi: 10.1016/j.fertnstert.2012.01.104. Epub 2012 Feb 2. PMID 22305103